CLINICAL TRIAL: NCT06636344
Title: Impact of Optimized Recruitment and Follow-up of Patients with Pseudoxanthoma Elasticum (PXE) by the PXE Reference Center At the CHU in Angers, France, Thanks to the Implementation of Alternating Pathways, Adapted to Age and Symptomatology, and Including Teleconsultations
Brief Title: Impact of Optimized Recruitment and Follow-up of Patients with Pseudoxanthoma Elasticum (PXE)
Acronym: REMOTE-PXE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC23_0305
Record Dates: First submitted 2024-10-02; First posted 2024-10-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Pseudoxanthoma Elasticum
MeSH Terms: conditions — Pseudoxanthoma Elasticum | interventions — ABCC6 protein, human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Pseudoxanthoma Elasticum — Answer to the PSQ-18, patient care confidence score (likert scale) and SF-12 questionaries at each visit, for an estimated duration of 15 minutes.

SUMMARY:
Pseudoxanthoma elasticum (PXE) is a rare genetic disorder characterized by ectopic calcifications in the skin, retina and arterial walls. Angers University Hospital is the national rare disease reference center (CRMR) for PXE. Although PXE is hereditary, its main clinical manifestations (unsightly skin lesions, intermittent arterial claudication, stroke, retinal bleeding and blindness) are delayed and slowly progress over the course of a lifetime. They are rarely life-threatening but have a major functional impact. To date, management of PXE is purely preventive and symptomatic. Three successive "states" can be individualized during PXE course, corresponding to three very different patient profiles in terms of age, clinical manifestations, occurrence of complications and their treatment.

PXE is essentially a severe disease in adults in the second half of life. This contrasts with the presence of many patients seen for their follow-up at school age or in employment, and at the age of children. It is therefore necessary to optimize the recruitment of PXE patients and to rethink their follow-up by the CRMR.

The investigators hypothesize that the implementation of alternating treatment paths, better adapted to each of the three patient profiles, including multidisciplinary teleconsultations, will not only increase the number of patients monitored by the CRMR and benefit from referral care, but also to optimize care, for greater patient satisfaction, their local doctors and the CRMR team.

DETAILED DESCRIPTION:
This is a quasi-experimental study evaluating the impact of new support modalities according to a before/after design with an intermediate transition period of 2 years necessary for the proper deployment of these new modalities. The study includes 3 separate periods of 2 years from its implementation:

* Period A1-2: continuation of the recruitment, monitoring and care methods for PXE patients as they are currently carried out. This period will allow the collection of baseline evaluation criteria
* Period A3-4 (intermediate period without evaluation/monitoring of indicators): gradual implementation of the internal organizational changes necessary for the deployment of alternating pathways.
* Period A5-6 (second period of interest for the evaluation of indicators): evaluation of fully operational alternating pathways for the recruitment, monitoring and care of PXE patients. This period will allow the collection of evaluation criteria and comparison with those of baseline).

For the main objective and the first secondary objectives relating to the optimization of the care pathway, the analysis will be carried out using global activity data at the CRMR level (non-identifying aggregated data).

This research involving humans is qualified as non-interventional research because to respond to :

* the second secondary objective about 'Evaluation of the impact of alternating courses adapted to age and clinical symptoms on the following criteria', patients will answer questionnaires specific to the study (quality of life, satisfaction and confidence for the patient and the treating physicians involved)
* the third secondary objective, semi-directed interviews will be carried out for patients, relatives (except parents) and treating physicians who agree to participate in the qualitative sub-study.

The overall activity data of the CRMR will be collected retrospectively and prospectively on the basis of all source data in order to characterize the evolution of the active file in terms of patients "duly followed up", "contacts without follow-up" or "lost to follow-up" during periods A1-A2 and A5-A6.

ELIGIBILITY:
Inclusion Criteria:

* For the main objective and the first secondary objectives : The population taken into account corresponds to all the support and requests managed by the CRMR over the periods of interest (period A1-2 and period A5-6).
* Inclusion in REMOTE-PXE is offered to any patient with a PXE, defined phenotypically or genotypically (see below), treated at the CRMR during the periods of interest. Note that inclusions are independent between the 2 periods (a patient included during period A1-2 can be included again if he/she is treated during period A5-6). PXE is defined phenotypically:
* by the presence of specific skin lesions (clinically suggestive and showing dermal elastorrhexis on skin biopsy) in patients under 25 years of age
* OR by the combination of specific skin lesions (clinically suggestive and showing dermal elastorrhexis on skin biopsy) and specific ophthalmologic lesions, complicated or not (depending on age: orange peel, angioid streaks, retinal dystrophy) over 25 years of age PXE is defined genotypically, regardless of the patient's age, by the identification of two variants in the ABCC6 gene.
* Participation in the qualitative study (semi-directed interviews) will be offered to a sample of patients included in the RIPH during the A5-A6 period among patients who were already followed before the A3-A4 period since the objective is to collect their experiences and perceptions of this reorganization of care. Only patients agreeing to participate in this sub-study and giving their consent for the recording of the interviews will be included.

Exclusion Criteria:

* Person objecting to participating in the research
* Patient under curatorship, guardianship and legal protection

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients belonging to the CRMR active cohort will be defined by:
  * for new patients: patients for whom CRMR care has been provided, i.e. a stay at the CRMR (consultation or hospitalization) or a teleconsultation with the CRMR team) was provided within a maximum of 3 months after an initial contact made during the period of interest
  * for patients already in the CRMR active file (patients who have benefited from at least one care in the last 5 years): patients for whom the CRMR care provided for the period, i.e. a stay at the CRMR (consultation or hospitalization) or a teleconsultation with the CRMR multidisciplinary team, was provided in accordance with the planned frequency with a tolerance window of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of alternating pathways adapted to age and clinical symptoms on the number of patients duly followed up | Patients duly followed correspond to: - New patients - Patient already followed at the CRMR corresponding to patients who have received at least one follow-up in the last 5 years whose this follow-up was carried out correctly in accordance with the plan
  Difference between the number of PXE patients duly followed up over the 2-year period (A5-6), after a period of implementation (2 years) of alternating pathways adapted to age, and the number of PXE patients duly followed up over the 2-year period following the implementation of the study (A1-2).

SECONDARY OUTCOMES:
Optimization of the care pathway by evaluating the impact of alternating pathways adapted to age and clinical symptoms | Comparison between the periode A5-6 (years 5 and 6) and A1-2 (years 1 and 2)
  The number of patients contacted without follow-up: Difference between the number of patients contacted without follow-up: during the period A5-6 and the period A1-2 The number of patients lost to follow-up: Difference between the number of patients lost to follow-up during the period A5-6 and the period A1-2 The time taken to take charge of new patients: Difference between the average time taken to the first effective care (face-to-face consultation, hospitalization or teleconsultation) and the first contact made during the period A1-2 and the period A5-6
Improving the quality of care by evaluating the impact of alternating pathways adapted to age and clinical symptoms on the following criteria | Comparison between the periode A5-6 (years 5 and 6) and A1-2 (years 1 and 2)
  The percentage of patients followed up with a new serious complication between period A5-6 and period A1-2
Improving the quality of care by evaluating the impact of alternating pathways adapted to age and clinical symptoms on the following criteria | Comparison between the periode A5-6 (years 5 and 6) and A1-2 (years 1 and 2)
  The number of patients followed up who completed all the necessary and prescribed examinations between period A5-6 and period A1-2
Improving the quality of care by evaluating the impact of alternating pathways adapted to age and clinical symptoms on the following criteria | Comparison between the periode A5-6 (years 5 and 6) and A1-2 (years 1 and 2)
  The satisfaction score relating to patient care between period A5-6 and period A1-2 using the short version of the PSQ (PSQ-18), a questionnaire regularly used to assess the relevance of telemedicine
  The PSQ-18 consisted of 18 statements including seven dimensions of satisfaction of medical care measured by : General Satisfaction; Technical Quality; Interpersonal Manner; Communication; Financial Aspects; Time Spent with Doctor; Accessibility and Convenience. Response were given on a five point scale ranging from strongly agree to strongly disagree. High scores reflect satisfaction with medical care
Improving the quality of care by evaluating the impact of alternating pathways adapted to age and clinical symptoms on the following criteria | Comparison between the periode A5-6 (years 5 and 6) and A1-2 (years 1 and 2)
  The confidence score relating to patient care between period A5-6 and period A1-2 (Likert scale from 0-Not at all confident to 5-Completely confident) assessed in patients and their treating physicians
Improving the quality of care by evaluating the impact of alternating pathways adapted to age and clinical symptoms on the following criteria | At enrollment and during routine case follow up (time frame is patient dependent)
  The quality of life score of patients between period A5-6 and period A1-2 using the SF-12 SF-12 : consists of 12 questions covering physical and mental health domains. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health
Improving the quality of care by evaluating the impact of alternating pathways adapted to age and clinical symptoms on the following criteria | At enrollment and during routine case follow up (time frame is patient dependent)
  The satisfaction score of the treating physician relating to patient care between period A5-6 and period A1-2 using the questionnaire SAPHORA.
  Calculation of a score per item: assignment of a scale to each modality of response whose value increases with the level of satisfaction (0-25-50-75-100)
Evaluation of the implementation of new alternating care pathways | 1 hour
  Semi-directed interviews will be carried out with the various stakeholders involved in this reorganization of care

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic Martin, Professor, Principal Investigator — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: No